CLINICAL TRIAL: NCT05290077
Title: Role of Serum NGAL Inearly Detection of CVR in Patients With Vitiligo
Brief Title: Role of NGAL in Vitiligo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Doaa Gamal Hafez, resident doctor at dermatology department sohag university hospital, Sohag University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Soh-Med-21-10-20
Record Dates: First submitted 2021-11-07; First posted 2022-03-22 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2021-12

CONDITIONS: Vitiligo
Keywords: NGAL & CVR
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cases (Active Comparator): group of vitiligo patients
  Interventions: Diagnostic Test: NGAL
- control group (Active Comparator): healthy group
  Interventions: Diagnostic Test: NGAL

INTERVENTIONS:
Diagnostic Test: NGAL — Serum NGAL in blood for early detection of CVR

SUMMARY:
Role of serum Neutrophil Gelatinase-associated Lipocalin in early detection of cardiovascular risk in patients with Vitiligo

ELIGIBILITY:
Inclusion Criteria:

* patients with vitiligo above 20y

Exclusion Criteria:

* patients with systemic disease Pregnants female Lactating females Patients less than 20 y Patients with active lesions

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2022-12-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
serum Neutrophil Gelatinase-associated Lipocalin in patients with Vitilig | 6 months
  Role of serum Neutrophil Gelatinase-associated Lipocalin in early detection of cardiovascular risk in patients with Vitiligo

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag fuculty, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ezzedine K, Eleftheriadou V, Whitton M, van Geel N. Vitiligo. Lancet. 2015 Jul 4;386(9988):74-84. doi: 10.1016/S0140-6736(14)60763-7. Epub 2015 Jan 15. PMID 25596811
- [Background] Vachiramon V, Onprasert W, Harnchoowong S, Chanprapaph K. Prevalence and Clinical Characteristics of Itch in Vitiligo and Its Clinical Significance. Biomed Res Int. 2017;2017:5617838. doi: 10.1155/2017/5617838. Epub 2017 Jul 30. PMID 28828385
- [Background] Silverberg JI, Silverberg NB. Association between vitiligo extent and distribution and quality-of-life impairment. JAMA Dermatol. 2013 Feb;149(2):159-64. doi: 10.1001/jamadermatol.2013.927. PMID 23560296
- [Background] Mazzei Weiss ME. Vitiligo: to biopsy or not to biopsy? Cutis. 2020 Apr;105(4):189-190. No abstract available. PMID 32463851